CLINICAL TRIAL: NCT05612529
Title: Ultrasonographic Predictors of Intravenous Fluid Responsiveness in Septic Shock and Its Correlation to Central Venous Pressure
Brief Title: Fluid Responseveness in Sepsis and Its Correlation to CVP
Status: Terminated | Type: Observational
Why Stopped: increase mortality rate in cases that made it difficult to follow up
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tasneem Hassan Younes, Assistant lecturer, Assiut University
Other Study IDs: fluid responseveness in sepsis
Record Dates: First submitted 2021-10-27; First posted 2022-11-10 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: US , Echocardiography — * Carotid ultrasonography: Parameters will be measured by single blinded independent examiner using an ultrasound device. Baseline carotid FTc, ΔVpeak, will be measured.
  * Echocardiography: Stroke Volume will be measured by transthoracic echocardiography.
  * Renal and splenic Doppler resistivity index.
  * Inferior vena cava collapsibility and distensibility indices.
  * Central venous pressure estimation by central venous catheter, and central - Lung ultrasound for detection of lung congestion
  * Lung ultrasound for detection of lung congestion.

SUMMARY:
Introduction Aim of the work Patients and methods Type of study Exclusion criteria Statistical analysis Research ethics Reference

DETAILED DESCRIPTION:
Septic shock is a serious infectious condition characterized by low blood pressure and multiple organ damage. One of the traditional recommendations is to administer intravenous fluids as the first step to improve blood pressure(1).

However, studies have shown that not every patient benefits from aggressive intravenous hydration (2).

Previous studies have shown that certain parameters may correlate with volume status and others may not to correlate with patient volume status.

Hemodynamic parameters, such as stroke volume variation (SVV) and pleth variability index (PVI) may better predict fluid responsiveness. However, assessments of these parameters require invasive procedures and special monitoring equipment, which limits their clinical application (4).

Echocardiography has been widely adopted to diagnose and monitor cardiac dysfunction leading to hemodynamic instability, and shock pathophysiology in general.

However, the echocardiographic information on macro-hemodynamics is partial, especially as being indirect as concerns vascular tone, and not allowing any inference on end-organ perfusion (5).

Recently, ultrasonography for estimating volume status has been widely recommended because of its non-invasive nature, ease of acquisition, and reproducibility of measurements.

The inferior vena cava (IVC) is a compliant vessel whose size and shape vary with changes in CVP and intravascular volume. Therefore, sonographic measurement of the IVC represents an effective and non-invasive method of estimating CVP.

Respiratory variation in the IVC diameter was used as a guide for fluid therapy in septic shock in both spontaneous breathing and mechanically ventilated patients.

Moreover, the assessment of visceral end-organ perfusion by ultrasound, may offer insights into this facet of shock pathophysiology (5).

Among these ultrasound modalities, corrected flow time (FTc) measured in the carotid artery is a new approach for predicting fluid responsiveness that has shown promising results.

Therefore, although it is a dynamic index, it may be able to adequately evaluate volume status in spontaneously and mechanically breathing patients.

Aim of the work: 1- To evaluate whether carotid FTc as determined by Doppler ultrasound could be a predictor of fluid responsiveness in spontaneously breathing and mechanically ventilated patients.

2- To evaluate the predictive ability of ΔVpeak for fluid responsiveness in spontaneously breathing patients.

3- To detect changes of regional splanchnic hemodynamics by color Doppler resistive index, and its improvement after fluid administration.

4- To evaluate the predictive ability of IVC collapsibility and distensibility indices for fluid responsiveness in septic shock patients.

5- To compare between the predictive ability of the measured Ultrasonographic parameters and the CVP changes in response to intravenous fluid therapy in both spontaneously breathing and mechanically ventilated septic shock patients.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients age≥18-year-old; written consent will be obtained.
2. septic shocked patients show signs of acute circulatory failure at any time within the first 72 hours.

Exclusion Criteria:

1. Patients confirmed to have cardiogenic shock.
2. History of heart failure or patient known to have moderate to severe valvular heart disease, congenital heart disease.
3. The presence of carotid artery stenosis >50% , newly detected common carotid stenosis >50% during the study period.
4. Non-sinus rhythm.
5. Moderate to severe anemia.
6. Markedly increased intraabdominal pressure as abdominal compartment syndrome, pregnancy.
7. Medically diseased kidneys, ureteric obstruction peri-nephric collection.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: After recording these data, the patients will be administered a fluid challenge of a 500 mL fluid bolus of 0.9% normal saline over 10 min and then same haemodynamic parameters will be measured again.
  Fluid responsiveness is an increase of stroke volume of 10-15% by echocardiography, after the patient receives 500 ml of crystalloid over 10 min.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic predictors of intravenous fluid responsiveness in septic shock and its correlation to central venous pressure | Baseline
  To evaluate whether carotid FTc as determined by Doppler ultrasound could be a predictor of fluid responsiveness in spontaneously breathing and MV patients.
Evaluation the predictive ability of ΔVpeak for fluid responsiveness in spontaneously breathing patients. | Baseline
  To evaluate the predictive ability of ΔVpeak for fluid responsiveness in spontaneously breathing patients.
  and the ΔVpeak will be calculated as follows: (maximum peak velocity - minimum peak velocity)/[(maximum peak velocity + minimum peak velocity)/2] × 100
Detection changes of regional splanchnic hemodynamics by color Doppler resistive index, and its improvement after fluid administration. | Baseline
  To detect changes of regional splanchnic hemodynamics by color Doppler resistive index, and its improvement after fluid administration.
  Resistive index (RI): (peak systolic velocity - end-diastolic velocity) / peak systolic velocity. The normal range is 0.50-0.70.

CONTACTS AND LOCATIONS:
Overall Officials: olfat M elshinawy, professor, Principal Investigator — Assiut University; mohamed M abdelhady, professor, Principal Investigator — Assiut University; arafa M aboelhassan, Principal Investigator — Assiut University
Locations (1):
- Tasneem Hassan Younes, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy MM, Evans LE, Rhodes A. The Surviving Sepsis Campaign Bundle: 2018 update. Intensive Care Med. 2018 Jun;44(6):925-928. doi: 10.1007/s00134-018-5085-0. Epub 2018 Apr 19. No abstract available. PMID 29675566
- [Background] Vandervelden S, Malbrain ML. Initial resuscitation from severe sepsis: one size does not fit all. Anaesthesiol Intensive Ther. 2015;47 Spec No:s44-55. doi: 10.5603/AIT.a2015.0075. Epub 2015 Nov 18. PMID 26578400
- [Background] Lammi MR, Aiello B, Burg GT, Rehman T, Douglas IS, Wheeler AP, deBoisblanc BP; National Institutes of Health, National Heart, Lung, and Blood Institute ARDS Network Investigators. Response to fluid boluses in the fluid and catheter treatment trial. Chest. 2015 Oct;148(4):919-926. doi: 10.1378/chest.15-0445. PMID 26020673
- [Background] Hu B, Xiang H, Liang H, Yu L, Xu T, Yang JH, DU ZH, Li JG. Assessment effect of central venous pressure in fluid resuscitation in the patients with shock: a multi-center retrospective research. Chin Med J (Engl). 2013;126(10):1844-9. PMID 23673097
- [Background] Corradi F, Via G, Tavazzi G. What's new in ultrasound-based assessment of organ perfusion in the critically ill: expanding the bedside clinical monitoring window for hypoperfusion in shock. Intensive Care Med. 2020 Apr;46(4):775-779. doi: 10.1007/s00134-019-05791-y. Epub 2019 Oct 25. No abstract available. PMID 31654077
- [Background] Kim HJ, Choi YS, Kim SH, Lee W, Kwon JY, Kim DH. Predictability of preoperative carotid artery-corrected flow time for hypotension after spinal anaesthesia in patients undergoing caesarean section: A prospective observational study. Eur J Anaesthesiol. 2021 Apr 1;38(4):394-401. doi: 10.1097/EJA.0000000000001376. PMID 33122575